CLINICAL TRIAL: NCT04073979
Title: MATTERS II - Mistral Percutaneous Tricuspid Valve Repair FIM Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mitralix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-605
Record Dates: First submitted 2019-08-25; First posted 2019-08-29 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Tricuspid Valve Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mistral (Experimental): The Mistral is an investigational device intended for percutaneous trans-catheter repair in high risk for surgery individuals suffering from functional Tricuspid Regurgitation (TR).
  The device system is to be used only in accordance with the approved Investigational Plan on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.
  Interventions: Device: Mistral implantation

INTERVENTIONS:
Device: Mistral implantation — Mistral implant is implanted in the Tricuspid valve

SUMMARY:
The Mistral is an investigational device intended for percutaneous trans-catheter repair in high risk for surgery individuals suffering from functional Tricuspid Regurgitation (TR).

The device system is to be used only in accordance with the approved Investigational Plan on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.

DETAILED DESCRIPTION:
The study is designed to clinically demonstrate device acute safety and technical performance (Primary Endpoints) along with longer FU device safety and effectiveness evaluation (Secondary Endpoint).

The main objectives of the study are:

* Evaluate the Acute safety of the implanted Mistral device post procedure and at 30 day follow up period.
* Evaluate the long term Safety of the device.
* Demonstrate effectiveness of the Mistral device in reducing TR.

Primary endpoints:

* Safety: Acute safety. Rate of all SAEs including device related SAEs, all caused mortality, stroke, MI, cardiac tamponade, surgery for failed percutaneous repair and non-elective cardiovascular surgery to treat an adverse event. At discharge and 30 days.
* Performance: Mistral Implantation rate of technical success (defined as successful device implantation with grasped chords from at least two leaflets.).

Secondary endpoints:

* Safety: Safety at 3,6, 12 and 24 months. Rate of all SAEs including device related SAEs at 3, 6, 12 and 24 months.
* Effectiveness: TR reduction post-procedure, at discharge and 30 days, 3,6, 12 and 24 months. Improved NYHA class, 6MWTdistance and KCCQ (quality of life) at 30 days, 3,6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject has given signed study Informed Consent for participation prior to procedure.
* Subject is ≥ 18 years of age or legal age in host country
* Subject is willing and able to comply with all required follow-up evaluations
* Genders eligible for the study: Both genders
* Chronic functional tricuspid regurgitation (FTR) with a minimum of moderate tricuspid regurgitation;

  o Subjects with moderate TR: Only NYHA Class III or IV maybe considered for inclusion.
* Subjects with severe or greater TR: NYHA II, III, or IV may be considered for inclusion Subject has left ventricular ejection fraction (LVEF) >20 %
* Subject is of functional class 2 or more (NYHA)
* The subject is high risk to undergo TV surgery as assessed and consented by a cardiac surgeon and an interventional cardiologist at the site (center heart team), and according to ESC/EACTS guidelines on the management of valvular heart disease.
* Patients with Jugular and/or Femoral veins enabling catheterization with 12Fr catheters
* Life expectancy ≥ 1 year

Exclusion Criteria:

* Tricuspid Stenosis >mild
* Tricuspid Subvalvular calcification or calcification of the chordae.
* Subjects with Aortic and/or Mitral valve severe stenosis and/or severe regurgitation.
* Subjects with severe, uncontrolled hypertension.
* Subjects with previous tricuspid repair or replacement.
* Subjects, which need to undergo an emergency surgery.
* Subjects participating in another clinical investigation.
* Subject has a history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within the past 90 days.
* Subject has a history of a myocardial infarction (MI) in the past 90 days.
* Subject has had a percutaneous interventional, including coronary intervention (PCI), within the last 90 days before procedure.
* Subject has a history of, or has active endocarditis
* Subject has echocardiographic evidence of intra-cardiac mass, thrombus, vegetation or soft-mobile deposits
* Subject is in acute pulmonary edema.
* Subject has hemodynamic instability requiring inotropic or mechanical support.
* Subject has a known hypersensitivity or contraindication to anticoagulant or antiplatelet medication.
* Subject has renal insufficiency as evidenced by a serum Creatinine > 3.0mg/dL.
* Subject has ongoing infection or sepsis
* Subject has blood dyscrasias (leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy)
* Subject has an active peptic ulcer or has had gastrointestinal (GI) bleeding within the past 3 months prior to the index procedure
* Subject requires emergency surgery for any reason
* Subject has a known allergy to Nitinol alloys, 316L\304 stainless steel.
* Pregnant or lactating women.
* Patients being dependent upon the sponsor or upon the investigator or upon the investigational site.
* Subject has a known contrast media allergy
* Presence of high degree atrio-ventricular block (2nd or 3rd degree A-V block), or the presence of tri-fascicular block
* According to investigator on site the patient is suffering from a severe end stage disease (e.g. malignancy, severe pulmonary disease, liver disease, renal failure) and has a life expectancy of less than 1 year.
* Contraindication for treatment with dual antiplatelet therapy for at least 3 months
* Contraindication for TEE including trans-gastric views.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Acute safety, Rate of device related SAE | Until hospital discharge - up to 5 days post procedure day
  including device related mortality, stroke, MI, cardiac tamponade, surgery for failed percutaneous repair and non-elective cardiovascular surgery to treat an adverse event.
Acute safety: Rate of device related SAE | At 30 days post procedure
  including device related mortality, stroke, MI, cardiac tamponade, surgery for failed percutaneous repair and non-elective cardiovascular surgery to treat an adverse event.
Performance: Mistral Implantation rate of technical success | Procedure
  defined as successful device implantation with grasped chords from at least two leaflets.

SECONDARY OUTCOMES:
Safety: Rate of all SAEs | At 3 months post procedure
  including device related SAEs
Safety: Rate of all SAEs | At 6 months post procedure
  including device related SAEs
Safety: Rate of all SAEs | At 12 months post procedure
  including device related SAEs
Safety: Rate of all SAEs | At 24 months post procedure
  including device related SAEs
Effectiveness TR | Until hospital discharge - up to 5 days post procedure day
  TR reduction
Effectiveness TR | At 30 days post procedure
  TR reduction
Effectiveness TR | At 3 months post procedure
  TR reduction
Effectiveness TR | At 6 months post procedure
  TR reduction
Effectiveness TR | At 12 months post procedure
  TR reduction
Effectiveness TR | At 24 months post procedure
  TR reduction
Effectiveness NYHA class | At 30 days post procedure
  Improved NYHA class (quality of life)
Effectiveness NYHA class | At 3 months post procedure
  Improved NYHA class (quality of life)
Effectiveness NYHA class | At 6 months post procedure
  Improved NYHA class (quality of life)
Effectiveness NYHA class | At 12 months post procedure
  Improved NYHA class (quality of life)
Effectiveness NYHA class | At 24 months post procedure
  Improved NYHA class (quality of life)
Effectiveness 6MWT | At 30 days post procedure
  Improved 6MWT distance (quality of life)
Effectiveness 6MWT | At 3 months post procedure
  Improved 6MWT distance (quality of life)
Effectiveness 6MWT | At 6 months post procedure
  Improved 6MWT distance (quality of life)
Effectiveness 6MWT | At 12 months post procedure
  Improved 6MWT distance (quality of life)
Effectiveness 6MWT | At 24 months post procedure
  Improved 6MWT distance (quality of life)
Effectiveness KCCQ | At 30 days post procedure
  Improved KCCQ (quality of life)
Effectiveness KCCQ | At 3 months post procedure
  Improved KCCQ (quality of life)
Effectiveness KCCQ | At 6 months post procedure
  Improved KCCQ (quality of life)
Effectiveness KCCQ | At 12 months post procedure
  Improved KCCQ (quality of life)
Effectiveness KCCQ | At 24 months post procedure
  Improved KCCQ (quality of life)

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Cardiovascular Center (CVC), Frankfurt
  - Marienkrankenhaus, Hamburg
  - Medizinisches Versorgungszentrum Albertinen (MVZ), Hamburg
  - LMU [Ludwig-Maximilians-Universität München], Munich